CLINICAL TRIAL: NCT06944678
Title: OHANA Project: Optimizing Health Care Through Alignment and Care Across Cultures
Brief Title: OHANA: Optimizing Cross-Cultural Care
Acronym: OHANA
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: Project OHANA - ID 7512
Record Dates: First submitted 2025-04-04; First posted 2025-04-25 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Cultural Competence

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Increasing globalisation and international migration have led to greater cultural diversity in Western societies, including healthcare settings. Hospitals and healthcare environments have become meeting places for individuals from different cultural backgrounds.

This diversity presents significant opportunities for improving healthcare, but also introduces complex challenges related to communication, trust and mutual understanding between healthcare professionals and patients. In this context, the concept of culturally competent care, i.e. the ability of healthcare professionals to provide respectful and appropriate care to patients by taking into account their cultural beliefs, values and practices, emerges as a crucial approach to address the specific needs of patients from different cultures. The concept of cultural competence was first introduced by Cross, who defines it as a set of behaviours, attitudes and policies that, when integrated into an organisation or among professionals, enable them to operate effectively in intercultural contexts.

DETAILED DESCRIPTION:
Although there is preliminary evidence on the benefits of cultural concordance, the literature is still scarce and fragmented. In particular, there is a lack of in-depth studies on the subjective experiences of the main actors involved. For healthcare professionals, cultural concordance could be a valuable resource, but also a source of additional stress or pressure, especially if perceived as a task requiring cultural or linguistic competence that is not always adequately supported. For patients, the experience of being cared for by a professional from the same culture might enhance a sense of trust and comfort, but also generate unrealistic expectations or influence perceptions of quality of care. Exploring the lived experiences of healthcare professionals and patients in a context of cultural concordance is essential to understanding perceived benefits, criticisms and areas for improvement. This multicentre study, coordinated by the Gemelli Hospital in Italy in collaboration with several Italian hospitals , aims to explore cultural concordance in a variety of healthcare settings, providing an in-depth understanding of the potentials and criticisms of cultural concordance in hospital settings

ELIGIBILITY:
Inclusion Criteria:

* All nurses or caregivers involved in the concordance system cultural will be included, with direct experience in caring for foreign patients
* All foreign patients admitted to hospital who speak a language other than the main language of the host country and who have been involved in the concordance system cultural will be included

Exclusion Criteria:

* All patients with severe cognitive conditions that prevent participation and nurses or caregivers who do not work closely with assigned patients will be excluded.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study will be conducted by enrolling participants who adopt a cultural concordance system.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Health workers' perceived utility of the cultural concordance system | 12 months
  Assessed through thematic content analysis of semi-structured interviews.
Socio-demographic characteristics of health workers | 12 months
  Collected using a socio-demographic questionnaire.

SECONDARY OUTCOMES:
Patients' perceptions of the cultural sensitivity of care received | 24 months
  Assessed through thematic content analysis of semi-structured interviews.
Socio-demographic characteristics of patients | 24 months
  Collected using a socio-demographic questionnaire.
Barriers to implementation of the cultural concordance system | 24 months
  Assessed through thematic content analysis of semi-structured interviews with health workers.
Facilitators to implementation of the cultural concordance system | 24 months
  Assessed through thematic content analysis of semi-structured interviews with health workers.
Development of evidence-based recommendations to improve cultural concordance | 24 months
  Number and content of guidelines produced based on interview data.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Pistacchio, PI, Principal Investigator — Fondazione Policlinico A. Gemelli IRCCS, Rome
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy